CLINICAL TRIAL: NCT04960319
Title: Prospective, ranDomized, Controlled, multicEnter Study for the Treatment of CALCIFied Coronary Artery Lesions With Rotational Atherectomy vs Intravascular LithotripsY
Brief Title: Rotablation vs Intravascular Lithotripsy in Calcified Coronary Lesions
Acronym: DECALCIFY
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Medical Care Center Prof. Mathey, Prof. Schofer, Ltd. (Other)
Collaborators: Shockwave Medical, Inc. (Industry); Asklepios proresearch (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DECALCIFY
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Coronary Artery Disease; Calcification
Keywords: Intravascular Lithotripsy; Rotational Atherectomy
MeSH Terms: conditions — Coronary Artery Disease; Calcinosis

STUDY DESIGN:
Intervention Model Description: Prospective, 1:1 randomized, controlled, multicenter trial to assess effectiveness and safety of Intravascular Lithotripsy (IVL) compared to Rotational Atherectomy (RA) treatment in calcified coronary lesions. An interim analysis after enrollment of 50 patients randomized will be performed. Based on the result the sample size will be calculated.
Who Masked: Outcomes Assessor
Masking Description: Core Lab is blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Intravascular Lithotripsy (Experimental): Study Device Treatment: IVL balloon catheter size is chosen in a 1:1 ratio to the distal reference vessel diameter. If the IVL balloon cannot be delivered into the target lesion a Guide catheter extension is recommended. The balloon catheter is then inflated to 4 ATM and 10 impulses are delivered. The balloon is then inflated to 6 ATM and deflated to reestablish blood flow. Up to 80 impulses can subsequently be delivered and the balloon can be repositioned within the lesion. In multiple lesions with different reference vessel diameters different sizes of IVL balloon can be used.
  Interventions: Device: Intravascular Lithotripsy
- Rotational Atherectomy (Active Comparator): Control group treatment: Rotablation should be performed as described in the ESC-Consensus document. Burr/vessel-ratio is 0.5 - 0.75. The use of different burr sizes as well as the use of a temporary pacemaker is left to the operator's discretion.
  Interventions: Device: Intravascular Lithotripsy

INTERVENTIONS:
Device: Intravascular Lithotripsy — Coronary Angiography. When the anatomic inclusion criteria are met, traverse the lesion with a guidewire. If traversal fails, assign the subject to the registry. After wire traversal has been documented by cine angiography, angiographic, OCT-defined or balloon expansion criteria are met, subject is enrolled. Blood sample for Troponin (hs TnT) baseline measurement has to be taken. The subjects will be randomized in a 1:1 fashion to treatment with either IVL or RA.

SUMMARY:
Prospective, 1:1 randomized, controlled, multicenter trial to assess effectiveness and safety of Intravascular Lithotripsy (IVL) compared to Rotational Atherectomy (RA) treatment in calcified coronary lesions

DETAILED DESCRIPTION:
1. Introduction

   Calcified coronary lesions are frequently observed and with increasing age and comorbidities of the patients they become even more prevalent (1,2). Calcified lesions are often difficult to dilate by conventional angioplasty leading to vessel perforation, dissection, or stent under-expansion, which impact survival, myocardial infarction rates, and target lesion revascularization (3 - 6). Lesion preparation before stent implantation has been strongly recommended using high-pressure dilatation, scoring/cutting balloons, or rotational atherectomy (RA) devices (7-12).

   RA can effectively modify calcified plaques by differential cutting, facilitating balloon dilatation, plaque fracture, stent delivery, and expansion (11). Patients undergoing RA experienced various clinical and angiographic complications, including vasospasm, perforation, short term vessel closure, side branch loss, and slow-flow/no-reflow resulting in stroke, myocardial infarction, and death (12). In the PREPARE-CALC trial (The Comparison of Strategies to Prepare Severely Calcified Coronary Lesions Trial) comparing RA and scoring or cutting balloons before drug-eluting stent implantation achieved a higher procedural success in RA (98% versus 81%), complications including larger dissection, perforation, and pericardial effusion were seen in 3%, 4%, and 3% of cases, respectively, in-hospital MACE occurred in 2% of cases (13). In the ORBIT II trial (14) an alternative atherectomy device was used which is based on the same mechanism of action as RA. In this trial the primary effectiveness performance goal, defined as successful stent delivery with residual stenosis < 50% and without in-hospital MACE, was not achieved in 11.1 % and the in-hospital MACCE rate was at 9.8 %, the rate of periprocedural myocardial infarction (MI), defined as CK-MB level > 3x ULN at discharge was 9.3% (non-Q-wave MI of 8.6 % and Q-wave MI of 0.7 %). Peri-procedural MI based on the 4th Universal Definition (15) after RA or ORBIT atherectomy have not been reported so far.

   Intravascular lithotripsy (IVL) disrupts subendothelial calcification by electrohydraulic-generated sonic pressure waves (16,17). In a recently published multicenter registry 78 patients were assigned to primary IVL therapy for patients with calcified de-novo lesions (n=39 lesions), secondary IVL therapy for patients with calcified lesions in which non-compliant balloon dilatation failed (n=22 lesions), and tertiary IVL therapy in patients with stent under expansion after previous stenting (n=17 lesions). The primary endpoint of strategy success (stent expansion with <20% in-stent residual stenosis) was reached in 84.6% with de-novo lesions with only 3 Type B dissections and no in-hospital MACCE (18). Recently Intravascular Lithotripsy for Treatment of Severely Calcified Coronary Artery Disease (Disrupt CAD III) Study (19) has been presented using the same in- and exclusion criteria as the ORBIT II study. The performance of IVL was compared with the performance of the ORBIT device, as being reported in the literature (14). The primary safety endpoint (cardiac death, or myocardial infarction, or target vessel revascularization) as well as the primary effectiveness endpoint (successful stent delivery with residual stenosis < 50 % and without in-hospital MACE) were 92.2 %, which were non-inferior to those reported in the ORBIT II study. Stent expansion was measured by QCA, data on OCT-based measurements of stent expansion in comparison to RA is not available. The rate of in-hospital peri-procedural MI, defined as CK-MB level > 3x ULN at discharge, was 6.8 %. Peri-procedural myocardial infarction and injury are associated with an increased rate of cardiovascular events at 30 days in patients undergoing elective coronary stenting (20).

   In order to evaluate the effectiveness of IVL in comparison to RA based on OCT- measurements of stent expansion and to study the incidence of in-hospital MACCE following either RA or IVL, we aim to perform a randomized trial.
2. Device Description and Intended Use

   Devices used in this study are commercially available and should be used according to labeled indications and the Manufacturers' Instructions for Use (IFU). Reference each device's IFU for a summary of the necessary training and experience needed to use the device and a description of the procedures involved in the use of the device.

   2.1. Intravascular Lithotripsy System

   The Intravascular Lithotripsy System (Shockwave Medical, Inc., Santa Clara, CA) is designed for the treatment of calcified coronary and peripheral artery stenosis. It is made up of three components: a battery-powered rechargeable generator capable of producing 3 kV energy and preprogramed to deliver a fixed number of pulses per balloon, a cable connector that links the generator with the catheter and a single-use sterile catheter with a semi-compliant balloon and three miniaturized lithotripsy emitters distributed along the length of the balloon. These emitters convert electrical energy into transient acoustic pressure pulses (1 pulse/s for a maximum of 80 pulses per catheter). IVL balloons are available in sizes ranging from 2.5 to 4.0 mm, with a unique maximum length of 12 mm. After the lithotripsy balloon is inflated to 405 kPa, pulsatile energy is emitted for 10 seconds from two emitters localized within the balloon (the distal emitter is slightly more central to enhance flexibility, whereas the proximal emitter is located near the proximal end of the balloon); the balloon is then inflated to 608 kPa. These balloons are compatible with 5 and 6 Fr guide catheters but have a rather large crossing profile of 0.043-0.046 inches. Detailed information can be found in the device related IFU.

   2.2. RotablatorTM Rotational Atherectomy System

   The RotablatorTM Rotational Atherectomy System (Boston Scientific Corp, MA) is designed for the treatment of calcified coronary artery lesions. It is made up of three components: a nickel-plated elliptic burr coated with diamond microscopic crystals that is available in sizes ranging from 1.25 to 2.50 mm diameter; a single advancer that can transmit rotational speed to the burr and is connected with a gas-driven turbine; and a control console and foot pedal. An ultrathin (0.009 inch) steerable dedicated guidewire (RotaWire) of length 330 mm is used to cross the calcified lesion; it is available in a floppy version or an extra support version, useful primarily in the treatment of aorto-ostial lesions. The RotaWire must be placed in the main vessel and other guidewires have to be removed from side branches to avoid wire cutting or perforation. When the burr is proximal to the lesion, rotablation can be started with short burr runs (<20 seconds) at a rotational speed of 135.000-180.000 rpm. A burr-to-artery ratio = 0.5-0.75 is adequate in most lesions as an initial approach, but occasionally it may be necessary to increase the burr size with a step-up approach. Fluoroscopic, acoustic and tactile signals should be monitored to avoid significant deceleration in rotational speed (>5,000 rpm), which is associated with complications.

   Detailed information can be found in the device related IFU.
3. Objectives

The objective of this prospective, 1:1 randomized, controlled, multicenter trial is to assess effectiveness and safety of Intravascular Lithotripsy (IVL) compared to Rotational Atherectomy (RA) treatment in calcified coronary lesions.

ELIGIBILITY:
Inclusion Criteria:

* Subject age ≥ 18 years
* Subject has been informed of the nature of the study, agrees to participate and has signed a Medical Ethics Committee approved consent form, understands the duration of the study, agrees to attend follow-up visits
* LVEF >25%
* Single de-novo target lesion with stenosis ≥ 70% and < 100% or ≥ 50% and < 70% with evidence of ischemia, or FFR ≤ 0.80, or lumen area ≤ 4.0 mm2 (≤ by 6.0mm2 in left main) IVUS or OCT
* Target vessel RVD ≥ 2.5 mm and ≤4.0 mm
* Lesion length ≤ 60 mm
* Lesion site severe calcification: Angiographic radio-opacities prior to contrast involving both sides of arterial wall with total calcium length ≥10 mm, or presence of ≥270° of calcium on at least one cross section by IVUS or OCT or incomplete balloon expansion at 12 atm
* Target lesion was traversed by a guide wire

Exclusion Criteria:

* Failure to successfully cross the target lesion with the guidewire
* Target lesion in a coronary artery bypass graft
* In-stent-Restenosis
* Thrombus in the target vessel
* Chronic total occlusion in the target vessel
* ST-elevation myocardial infarction (STEMI) within the last 4 weeks prior to enrollment
* Stroke within the last 3 months prior to enrollment
* Decompensated heart failure
* Life expectancy of less than one year
* Chronic kidney disease (serum creatinine > 2.5mg/dl)
* Pregnant or lactating females
* Receiving dialysis or immunosuppressant therapy
* Platelet Count < 100.000mm3 or > 600.000mm3
* Significant gastrointestinal bleeding or any coagulopathy that would contraindicate the use of antiplatelet therapy
* Known allergies or sensitivity to heparin, aspirin, other anticoagulant/antiplatelet therapies or contrast media that cannot be adequately pre-treated prior to index procedure
* Surgical procedure within the last 30 days prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Percent of stent expansion evaluated by Optical Coherence Tomography assessed by core lab. | at the end of the intervention
  Primary Effectiveness endpoint
Rate of in-hospital MACCE | 72 hours
  primary Safety endpoint

SECONDARY OUTCOMES:
Percentage of mean stent expansion evaluated by optical coherence tomography as assessed by core lab. | at the end of the intervention
  Secondary Effectiveness Endpoint
Rate of peri-procedural myocardial injury ,Peri-procedural myocardial infarction, Slow flow/no-reflow | 72 hours
  secondary safety endpoints

CONTACTS AND LOCATIONS:
Overall Officials: Joachim Schofer, MD, PhD, Principal Investigator — Medical Care Center Prof. Mathey, Prof. Schofer

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: at the time of publication